CLINICAL TRIAL: NCT06108609
Title: Validation of the French Version of the Hearing Aid Benefit Measurement COSI and IOI-HA Questionnaires
Acronym: AUDI-FR
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MDL_2023_7
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hearing Impairment
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Administration of the French version of the COSI and IOI-HA questionnaires — Inclusion (D0):
  * Audiometry (as part of treatment)
  * Clinical evaluation (as part of treatment)
  * Passing the French version of the COSI and IOI-HA questionnaires Visit 1 (D0 +3±1 week): only for 35 patients Second administration of the French version of the COSI and IOI-HA questionnaires either by telephone, or during a second consultation or hospitalization, if this occurs within a compatible time frame.

SUMMARY:
Estimating patient satisfaction is essential in modern day-to-day medical practice. This is particularly true in the field of audiology where evaluating the benefit of patients' devices makes it possible to improve settings and increase patient satisfaction and therefore compliance. Questionnaires measuring hearing aid benefit such as the IOI-HA (International Outcome Inventory for Hearing Aids) and the COSI (Client Oriented Scale of Improvement) are used in everyday practice and promote cooperation between researchers by providing comparable data. Unlike other countries, these questionnaires have never been validated in French by psychometric studies. The objective of this study is to validate the translation of the IOI-HA questionnaire already used in the clinic and to adapt the COSI into French and statistically validate its translation.

DETAILED DESCRIPTION:
Recruitment of cases via the otological consultation of the ENT department, among patients consulting for hearing aids. Inclusion will be suspended once 100 tests and at least 35 re-tests have been completed.

Inclusion (D0):

* Audiometry (as part of treatment)
* Clinical evaluation (as part of treatment)
* Passing the French version of the COSI and IOI-HA questionnaires Visit 1 (D0 +3±1 week): only for 35 patients Second administration of the French version of the COSI and IOI-HA questionnaires either by telephone, or during a second consultation or hospitalization, if this occurs within a compatible time frame.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Diagnosis of deafness with unilateral or bilateral hearing aid
* Informed consent to participate in the study
* Good understanding of French
* Non-opposition to participation in the study

Exclusion Criteria:

* Comorbidity that may hamper the interpretation of results (e.g. disabling cognitive disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients seen for consultation, with unilateral or bilateral hearing aids
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Statistical validation of the French version of the IOI-HA and COSI questionnaires: Reproducibility, internal consistency, relevance and discriminatory performance of the tests | 3 +/- 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Fondation Adolphe de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No